CLINICAL TRIAL: NCT00365846
Title: "A Pilot Study to Determine the Safety of Campath-1H (Anti-CD52) Therapy in Primary Renal Allograft Transplantation
Brief Title: "A Pilot Study to Determine the Safety of Campath-1H (Anti-CD52) Therapy in Primary Renal Allograft Transplantation"
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2000-032
Record Dates: First submitted 2006-08-16; First posted 2006-08-18 (Estimated); Results first posted 2012-07-30 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-09

CONDITIONS: Renal Transplant
Keywords: prevent kidney rejection
MeSH Terms: interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Campath 1H induction w/ Sirolimus immunosuppression (Experimental): Campath 1H at day -1 and 0 of kidney transplant followed by long term CNI free immunosuppressive therapy with Sirolimus,
  Interventions: Drug: Campath-1H

INTERVENTIONS:
Drug: Campath-1H

SUMMARY:
The purpose of the study is to see if campath-1H can be used in first time renal transplant subjects to prevent rejection and reduce the overall amount of anti-rejection medications that patients take on a daily basis.

DETAILED DESCRIPTION:
Twenty nine primary recipients of either a live donor or deceased donor renal transplant were enrolled in this study. Subjects were administered two 20mg doses of Campath-1H antibody therapy (Day 0 and Day 1) in combination with a short course of corticosteroids, and maintenance sirolimus.

Subjects were followed for 3 years to compare the incidence and severity of rejection episodes, complications related to the immunosuppression, including infections, malignancies and adverse events. All subjects underwent protocol renal transplant biopsies at 6 and 12 months (unless medically contraindicated).

ELIGIBILITY:
Inclusion Criteria:

* primary renal transplant (not HLA identical)
* ages 18-60 years

Exclusion Criteria:

* recipient panel reactive antibody level >10%
* recipient of a DCD kidney
* no prior organ transplant
* no multi-organ transplant recipient
* no subject who is currently receiving systemic corticosteroids
* no pregnant or lactating subjects
* no history of Hepatitis B, C or HIV positivity
* no recipient of a kidney with cold ischemia time >36 hours

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2000-08; Primary Completion 2005-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J Knechtle, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Result] Barth RN, Janus CA, Lillesand CA, Radke NA, Pirsch JD, Becker BN, Fernandez LA, Thomas Chin L, Becker YT, Odorico JS, D'Alessandro AM, Sollinger HW, Knechtle SJ. Outcomes at 3 years of a prospective pilot study of Campath-1H and sirolimus immunosuppression for renal transplantation. Transpl Int. 2006 Nov;19(11):885-92. doi: 10.1111/j.1432-2277.2006.00388.x. PMID 17018123
- [Derived] Fehr T, Hubel K, de Rougemont O, Abela I, Gaspert A, Gungor T, Hauri M, Helmchen B, Linsenmeier C, Muller T, Nilsson J, Riesterer O, Scandling JD, Schanz U, Cippa PE. Successful Induction of Specific Immunological Tolerance by Combined Kidney and Hematopoietic Stem Cell Transplantation in HLA-Identical Siblings. Front Immunol. 2022 Jan 31;13:796456. doi: 10.3389/fimmu.2022.796456. eCollection 2022. PMID 35173720

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Campath 1H induction w/ Sirolimus immunosuppression
Period: Overall Study
Arm/Group | Group 1
Started | 29
Completed | 28
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Age Continuous [Mean (Full Range); unit: years] | 41 [19 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Allograft Rejection
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Group 1
Number analyzed (Participants) | 28
participants | 13

2. Secondary Outcome: Incidence of Severe Allograft Rejection ( Defined as >Banff 2A or Requiring Antibody Treatment)
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Group 1
Number analyzed (Participants) | 28
participants | 6

3. Secondary Outcome: Patient Survival
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Group 1
Number analyzed (Participants) | 28
participants | 28

4. Secondary Outcome: Incidence of Post-transplant Infection
Description: Event of post-transplant infection (more than one "event" might have been counted per participant)
Time Frame: 3 years
Measure: Number; unit: event of infection
Groups:
- Campath 1H Induction w/ Sirolimus Immunosuppression: Campath 1H induction on Day -1 and 0 of renal transplant followed w/ Sirolimus maintenance immunosuppression
Arm/Group | Campath 1H Induction w/ Sirolimus Immunosuppression
Number analyzed (Participants) | 28
event of infection | 28

5. Secondary Outcome: Incidence of Malignancies
Description: Number of Participants Experiencing Malignancies
Time Frame: 3 years
Measure: Number; unit: participants
Groups:
- Group 1Campath 1H Induction w/ Sirolimus Immunosuppression: Campath 1H induction w/ Sirolimus immunosuppression
Arm/Group | Group 1Campath 1H Induction w/ Sirolimus Immunosuppression
Number analyzed (Participants) | 28
participants | 2

6. Secondary Outcome: Kidney Allograft Survival
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Group 1
Number analyzed (Participants) | 28
participants | 27

ADVERSE EVENTS:
Time Frame: Reported Adverse Events include events starting on of after Day 0 (day of Transplant) and on or before Month 36.
Description: If a subject experienced more than 1 or a given AE, the subject is counted only once for that AE. If a subject experienced more than one AE in a system organ class (SOC), the subject is counted only once in that SOC
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 19/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=28)
Acute kidney graft rejection (Renal and urinary disorders) | 13 (24)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Congestive Heart Failure (Cardiac disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Fever of unknown origin (General disorders) | 2 (2)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1)
Herpes Zoster (Infections and infestations) | 3 (3)
Herpes simplex (Infections and infestations) | 5 (5)
Iliac artery stenosis (Vascular disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5)
Renal Hematoma (Renal and urinary disorders) | 1 (1)
Renal parenchyma leak (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 10 (15)
Vesico-ureteral reflux (Renal and urinary disorders) | 1 (1)
abdominal hernia (Musculoskeletal and connective tissue disorders) | 7 (8)
acute renal insufficiency (Renal and urinary disorders) | 2 (2)
basal cell skin cancer (Skin and subcutaneous tissue disorders) | 2 (2)
bilateral extremity weakness (Nervous system disorders) | 1 (1)
drug toxicity (Injury, poisoning and procedural complications) | 1 (1) — Prograf toxicity
hypocalcemia (General disorders) | 1 (1)
intra abdominal abcess (Musculoskeletal and connective tissue disorders) | 2 (2)
kidney graft failure (Renal and urinary disorders) | 1 (1)
lymphocele (Renal and urinary disorders) | 2 (2)
myocardial Infarction (Cardiac disorders) | 1 (1)
pyelonephritis (Renal and urinary disorders) | 1 (1)
right ankle fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
secondary hyperparathyroidism (Endocrine disorders) | 1 (1)
ureteral stricture (Renal and urinary disorders) | 1 (1)
urosepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Group 1 (N=28)
anemia (Blood and lymphatic system disorders) | 10 (10) — mild
hyperlipidemia (Endocrine disorders) | 19 (19)
hyperglysemia (Endocrine disorders) | 4 (4) — steroid induced
proteinuria (Renal and urinary disorders) | 5 (5)
leukopenia (Blood and lymphatic system disorders) | 5 (5)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 7 (7)
osteopenia (Musculoskeletal and connective tissue disorders) | 6 (6)
insomnia (Psychiatric disorders) | 3 (3)
laceration (Injury, poisoning and procedural complications) | 2 (2) — finger
cataracts (Eye disorders) | 2 (2)
sleep apnea (Ear and labyrinth disorders) | 2 (2)
erectile dysfunction (Reproductive system and breast disorders) | 4/19 (4)
elevated liver enzymes (Hepatobiliary disorders) | 7 (7)
edema (Musculoskeletal and connective tissue disorders) | 5 (5) — lower extremity
Gastroesophageal reflux (Gastrointestinal disorders) | 7 (7)
amenorrhea (Reproductive system and breast disorders) | 2/7 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No